CLINICAL TRIAL: NCT07332221
Title: Application of Toripalimab as Adjuvant Therapy After Esophageal Cancer Surgery: A Multicenter, Phase III Clinical Trial
Brief Title: Application of Toripalimab as Adjuvant Therapy After Esophageal Cancer Surgery: A Multicenter Clinical Trial
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, YanZheng,MD, Director of Clinical Trials Center, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-586
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ypN+，receive toripalimab monotherapy as maintenance treatment (Experimental): R0 resection for esophageal cancer, ypN+
  Interventions: Drug: Toripalimab monotherapy
- ypN-，receive toripalimab monotherapy as maintenance treatment (Experimental): R0 resection for esophageal cancer, ypN-，receive toripalimab monotherapy as maintenance treatment
  Interventions: Drug: Toripalimab monotherapy
- ypN-，clinical observation only (No Intervention): R0 resection for esophageal cancer, ypN-，no further treatment

INTERVENTIONS:
Drug: Toripalimab monotherapy — Toripalimab monotherapy as maintenance treatment
  Arms: ypN+，receive toripalimab monotherapy as maintenance treatment; ypN-，receive toripalimab monotherapy as maintenance treatment

SUMMARY:
This study is a prospective, multicenter, multi-cohort Phase III clinical trial. It primarily enrolls high-risk recurrent esophageal cancer patients who have undergone R0 resection after neoadjuvant chemoimmunotherapy. Eligible patients are stratified based on pathological lymph node status and receive either toripalimab monotherapy as maintenance treatment or clinical observation only.

DETAILED DESCRIPTION:
This is a prospective, multicenter, multi-cohort Phase III clinical study. It primarily enrolls high-risk recurrent esophageal cancer patients who have achieved R0 resection after undergoing neoadjuvant chemoimmunotherapy. Eligible patients are stratified into two cohorts based on pathological lymph node status: Cohort A (ypN+ cohort) and Cohort B (ypN0 cohort).

Interventions and Treatment Schedule Cohort A (ypN+ cohort): Patients receive toripalimab monotherapy as consolidation/maintenance treatment.

Dosage: Toripalimab 240 mg. Administration: Every 3 weeks per cycle. Duration: Up to 17 cycles, with a total treatment period not exceeding one year.

Cohort B (ypN0 cohort): Patients are randomized 1:1 into two groups:

Experimental Group: Receives toripalimab monotherapy as consolidation/maintenance treatment (same dosage and schedule as Cohort A).

Control Group: Undergoes postoperative observation only. Follow-up and Assessments Disease Evaluation: Assessments including chest + upper abdominal contrast-enhanced CT + neck contrast-enhanced CT are performed every 3 months for 2 years, then every 6 months until the 5th year. PET-CT, chest MRI, gastroscopy, and bronchoscopy are conducted when necessary.

Safety Monitoring: Adverse events (AEs) are monitored throughout the study and graded according to CTCAE v5.0. Safety follow-up is performed for all subjects who received the study treatment, including those who discontinued early.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in this study, sign the informed consent form, demonstrate good compliance, and cooperate with follow-up.
2. Initial patients are those with resectable or potentially resectable (T1 N1-3 M0 or T2-3 N0-3 M0) thoracic segment esophageal squamous cell carcinoma (8th UICC-TNM staging); who have undergone surgical resection after 2 cycles of immunotherapy combined with chemotherapy and achieved R0 resection.
3. Age 18 to 75 years.
4. Preoperative examinations of various organ functions indicate no surgical contraindications.
5. The following laboratory tests confirm that bone marrow, liver, and kidney functions meet the study requirements:

   Hemoglobin ≥ 90 g/L; White blood cell count ≥ 4.0 × 10⁹/L; Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L; Platelet count ≥ 100 × 10⁹/L; Total bilirubin ≤ 1.5 times the upper limit of normal (ULN); ALT and AST ≤ 2.5 times ULN; International normalized ratio (INR) of prothrombin time ≤ 1.5 times ULN, and activated partial thromboplastin time within the normal range; Creatinine ≤ 1.5 times ULN.
6. No postoperative chemotherapy, radiotherapy, or hormone therapy for malignant tumors has been administered; no history of other malignancies, excluding prostate cancer patients who have received hormone therapy and achieved disease-free survival (DFS) for over 5 years.
7. Physical status ECOG score 0 to 1.
8. Women of childbearing potential must agree to use contraceptive measures (e.g., intrauterine device, contraceptive pills, or condoms) during the study and for 6 months after study completion; serum or urine pregnancy test within 7 days before study enrollment must be negative, and patients must be non-lactating; men must agree to use contraceptive measures during the study and for 6 months after study completion.

Exclusion Criteria:

1. Patients with double primary cancers;
2. Patients with infections requiring treatment;
3. Patients requiring continuous systemic corticosteroid therapy (Note: Replacement therapy (e.g., for thyroid insufficiency, insulin therapy, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered systemic therapy and is permitted);
4. Patients with unstable angina within 3 months or myocardial infarction within 6 months;
5. Patients with psychiatric disorders;
6. Patients with existing or concurrent hemorrhagic disorders;
7. Female patients who are pregnant or breastfeeding;
8. Patients with bronchial asthma requiring intermittent use of bronchodilators or medical intervention;
9. Patients who have used immunosuppressive agents prior to enrollment due to comorbid conditions, with a dose equivalent to ≥10mg/day of oral prednisone sustained for more than 2 weeks;
10. Patients with abnormal coagulation function (PT > 16s, APTT > 53s, TT > 21s, Fib < 1.5g/L), bleeding tendency, or those receiving thrombolytic or anticoagulant therapy;
11. Patients with pre-existing or concurrent pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, severe pulmonary impairment, etc.;
12. Patients with autoimmune diseases, immunodeficiency, or organ transplantation;
13. Patients with active Hepatitis B or Hepatitis C infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2031-10-01 (Estimated)

PRIMARY OUTCOMES:
2-year OS | every 3 months for 2 years
  the percentage of patients in a study who are still alive after 2years

SECONDARY OUTCOMES:
DFS | every 6 months until the 5th year
  DFS is defined as the time from surgery to any of the following events: local or distant recurrence, or death for any reason
OS | every 6 months until the 5th year
  OS (Overall Survival) is defined as the time from randomization (or treatment initiation) to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zheng, M.D., Principal Investigator — Henan Cancer Hospital